CLINICAL TRIAL: NCT06952413
Title: An Exploratory, Placebo-controlled, Double-blind, Phase II Study of the Efficacy and Safety for Rituximab (Genetical Recombination) in Myalgia Encephalomyelitis/Chronic Fatigue Syndrome (ME/CFS)
Brief Title: Study of the Efficacy and Safety for Rituximab in Myalgia Encephalomyelitis/Chronic Fatigue Syndrome (ME/CFS)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Center of Neurology and Psychiatry, Japan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IDEC-C2B8-MC
Record Dates: First submitted 2025-04-09; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Myalgia Encephalomyelitis/Chronic Fatigue Syndrome (ME/CFS)
MeSH Terms: conditions — Fatigue Syndrome, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rituximab(Genetical Recombination) (Active Comparator)
  Interventions: Drug: Rituximab(Genetical Recombination)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rituximab(Genetical Recombination) — Subjects will be assigned to the rituximab pre-treatment group or placebo pre-treatment group and will receive the study drug (rituximab actual or rituximab placebo) intravenously four times at weekly intervals during the first three weeks of the primary and secondary evaluation periods.
  Arms: Rituximab(Genetical Recombination)
Drug: Placebo — Subjects will be assigned to the rituximab pre-treatment group or placebo pre-treatment group and will receive the study drug (rituximab actual or rituximab placebo) intravenously four times at weekly intervals during the first three weeks of the primary and secondary evaluation periods.
  Arms: Placebo

SUMMARY:
The efficacy and safety of rituximab on ME/CFS symptoms after administration to patients with myalgic encephalomyelitis/chronic fatigue syndrome will be compared in an exploratory, placebo-controlled, double-blind fashion. In the subsequent secondary evaluation period, subjects who received rituximab in the primary evaluation period will receive placebo, and the timing and duration of rituximab's effect will be explored throughout the entire evaluation period. Subjects who received placebo during the primary evaluation period will receive rituximab during the secondary evaluation period to explore changes in endpoints before and after switching from placebo to rituximab in the same subjects.

DETAILED DESCRIPTION:
The efficacy and safety of rituximab (genetical recombination), a CD20 antibody, on ME/CFS symptoms after administration to patients with myalgic encephalomyelitis/chronic fatigue syndrome will be compared in an exploratory, placebo-controlled, double-blind fashion. In the subsequent secondary evaluation period, subjects who received rituximab in the primary evaluation period will receive placebo, and the timing and duration of rituximab's effect will be explored throughout the entire evaluation period. Subjects who received placebo during the primary evaluation period will receive rituximab during the secondary evaluation period to explore changes in endpoints before and after switching from placebo to rituximab in the same subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with ME/CFS who meet the Canadian criteria by a physician.
2. Patients with a severity score of 4 or higher on the Performance Status (PS) based ME/CFS severity classification by the Ministry of Health, Labour and Welfare Research Group
3. Patients who are between 18 and 65 years of age at the time of obtaining written consent
4. Patients who can be hospitalized (hospitalized from the day before administration and discharged the day after administration) at the time of the first dose of each of the primary and secondary evaluation periods
5. Patients whose written consent has been obtained

Exclusion Criteria:

1. Patients with a history of severe hypersensitivity or anaphylactic reactions to components of rituximab or products derived from mouse protein
2. Patients whose cardiopulmonary function is judged by the treating physician to be not maintained
3. Patients complaining of fatigue that does not meet the diagnostic criteria for ME/CFS
4. Patients found to have other medical conditions that may cause symptoms
5. Patients who are pregnant, lactating, or have a positive pregnancy test (serum human chorionic gonadotropin test) at the time of enrollment
6. Patients with coexisting or pre-existing malignant tumors (excluding basal cell carcinoma of the skin and cervical dysplasia)
7. Patients with coexisting or pre-existing severe immune system diseases (excluding autoimmune diseases such as thyroiditis and type 1 diabetes)
8. Patients with a history of systemic immunosuppressive therapy (e.g., immunoglobulin therapy, azathioprine, cyclosporine, mycophenolate mofetil, etc.) within 1 year, a history of receiving drugs such as monoclonal antibodies acting on the immune system (e.g., anti-CD20 antibody products including rituximab), or a history of comorbidities requiring treatment with immunosuppressive drugs Patients with comorbidities requiring treatment with immunosuppressive agents (excluding treatment with low-dose steroids of 5 mg /day or less)
9. Patients who have started alternative medicine (reference: acupuncture, moxibustion, and Japanese warm therapy) within 12 weeks prior to the start of treatment with the investigational drug.
10. Patients with severe endogenous (primary) depression
11. Patients with a neutrophil count <1.5*103/microliter and platelet count <10.0*104/microliter on blood test
12. Patients with impaired renal function (serum creatinine level > 1.5 times the upper limit of the reference value at the institution)
13. Patients with impaired hepatic function (serum bilirubin, Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT) levels exceeding 1.5 times the upper limit of the reference value of the institution)
14. Patients infected with Human Immunodeficiency Virus (HIV)
15. Patients who test positive for at least one of Hepatitis B surface (HBs) antigen, HBs antibody, Hepatitis B core (HBc) antibody, or Hepatitis C virus (HCV) antibody.

    However, patients who meet the following conditions (1) and (2) may be registered.

    (i) Patients who are positive for HBs or HBc antibodies and whose HBV-DNA quantification is confirmed to be negative (less than detection sensitivity) and for whom appropriate monitoring, etc. can be conducted in accordance with the Guidelines for Hepatitis B Treatment edited by the Japan Society of Hepatology.

    (ii) For patients with positive HCV antibody, when HCV-RNA quantification is negative (less than detection sensitivity)
16. Patients who do not have the ability to comply with the study protocol
17. Patients who have participated in other clinical trials or clinical studies (except for observational studies without intervention) within 16 weeks prior to obtaining consent
18. Other patients who are judged by the investigator or subinvestigator (hereinafter referred to as investigator) to be inappropriate to participate in this clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-09 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Improvement rate | From Baseline to the end of treatment at 24 weeks
  Percentage of cases in which the severity score of ME/CFS based on PS by the MHLW research group improved by 1 or more compared to that before the start of study drug administration (week 0)

SECONDARY OUTCOMES:
Percentage of patients whose MHLW-PS-based ME/CFS severity score improved by 1 or more at each evaluation point (improvement rate) compared to that before the start of treatment with the investigational drug (week 0). | At 4-week intervals from Baseline up to Week 48
The amount of change in the severity score of ME/CFS based on PS by the MHLW Research Group at each assessment point from that before the start of treatment with the investigational drug (week 0) | At 4-week intervals from Baseline up to Week 48
Proportion of awake time spent in supine position (%),Proportion of awake time spent in sitting position (%) | At 4-week intervals from Baseline up to Week 48
  Changes in proportions will be aggregated.
Duration of standing and activity (hours) | At 4-week intervals from Baseline up to Week 48
  Changes in time will be aggregated.
Fatigue during rest and lying position | At 4-week intervals from Baseline up to Week 48
  Patients will be asked to report the level of fatigue they feel even while lying down, and changes in their fatigue levels will be aggregated.
Records on exertion and Post-Exertional Malaise (PEM) | At 4-week intervals from Baseline up to Week 48
  Patients will be asked to describe the specific activities they perform and the exhaustion they experience afterward, and a summary table will be created.
Assessment of fatigue during physical activity | At 4-week intervals from Baseline up to Week 48
  Patients will be asked to report the level of fatigue they experience during physical activity in daily life, and changes in fatigue levels will be aggregated.
Evaluation based on Fatigue Score | At 2-week intervals from Baseline up to Week 48
  Patients will be asked to complete the Fatigue Score questionnaire, and changes in the score will be aggregated.
SF-36 | At 12-week intervals from Baseline up to Week 48
  Changes in scores obtained from the SF-36 questionnaire will be assessed to evaluate patients' quality of life.
COMPASS31 | At 12-week intervals from Baseline up to Week 48
  Changes in scores obtained from the COMPASS31 questionnaire will be assessed to evaluate patients' autonomic symptoms.
Pittsburgh Sleep Quality Index (PSQI) | At 12-week intervals from Baseline up to Week 48
  Changes in scores obtained from the PSQI questionnaire will be assessed to evaluate patients' sleep quality.
Pain intensity | At 12-week intervals from Baseline up to Week 48
  Pain intensity will be assessed using the Visual Analogue Scale (VAS)
Grip strength | At 12-week intervals from Baseline up to Week 48
  Patients' grip strength will be measured, and changes in the measurements will be aggregated.
Analysis of the gut microbiota | At 24-week intervals from Baseline up to Week 48
  samples collected from patients will be analyzed, and the composition of the gut microbiota will be aggregated.
Brain imaging evaluation (Magnetic Resonance Imaging (MRI) of the head, Single Photon Emission Computed Tomography (SPECT) of cerebral blood flow) | At 24-week intervals from Baseline up to Week 48
  Findings from imaging will be aggregated.
Immune biomarker analysis (qPCR) | At 24-week intervals from Baseline up to Week 48
  qPCR will be measured, and changes in their levels will be aggregated.
Immune biomarker analysis (anti-autonomic receptor antibody analysis) | At 24-week intervals from Baseline up to Week 48
  Quantify the level of anti-autonomic receptor antibodies will be measured, and changes in their levels will be aggregated.
Immune biomarker analysis (immune cell subfractionation analysis) | At 24-week intervals from Baseline up to Week 48
  The subsets of immune cells will be measured, and changes in the levels will be aggregated.
Metabolome analysis | At Baseline
  A detailed characterization of the patients' metabolome at baseline will be conducted.
Adverse events | From Baseline up to Week 48
  The number of adverse events will be aggregated.
Vital signs (body temperature) | Assessments will be conducted at baseline and at Weeks 1, 2, 3, 4, 8, 12, 24, 25, 26, 27, 28, 32, 36, and 48
  Summary statistics of vital signs will be calculated to monitor changes over time.
Vital signs (blood pressure) | Assessments will be conducted at baseline and at Weeks 1, 2, 3, 4, 8, 12, 24, 25, 26, 27, 28, 32, 36, and 48
  Summary statistics of vital signs will be calculated to monitor changes over time.
Vital signs (pulse rate) | Assessments will be conducted at baseline and at Weeks 1, 2, 3, 4, 8, 12, 24, 25, 26, 27, 28, 32, 36, and 48
  Summary statistics of vital signs will be calculated to monitor changes over time.
Serum immunoglobulins (IgG) | At 4-week intervals from Baseline up to Week 48
  Summary statistics of serum immunoglobulins will be calculated to monitor changes over time.
Serum immunoglobulins (IgM) | At 4-week intervals from Baseline up to Week 48
  Summary statistics of serum immunoglobulins will be calculated to monitor changes over time.
Serum immunoglobulins (IgA) | At 4-week intervals from Baseline up to Week 48
  Summary statistics of serum immunoglobulins will be calculated to monitor changes over time.
Rituximab concentration of the blood plasma | Assessments will be conducted at baseline and at Weeks 1, 2, 3, 4, 12, 24, 25, 26, 27, 28, 36, and 48
  Rituximab concentration of the blood plasma
Blood drug concentration Anti-Drug Antibody (ADA) | Assessments will be conducted at baseline and at Weeks 4, 12, 24, 28, 36, and 48.
  Summary statistics of ADA will be calculated to monitor changes over time.
B cells (CD19/CD20 positive cells) and T cells (CD3/CD4/CD8 positive cells) | Assessments will be conducted at baseline and at Weeks 1, 12, 24, 25, 36, and 48.
  Summary statistics of B cells and T cells will be calculated to monitor changes over time.

CONTACTS AND LOCATIONS:
Overall Officials: Tomoko Okamoto, MD, Principal Investigator — National Center of Neurology and Psychiatry
Locations (1):
- National Center of Neurology and Psychiatry, Kodaira, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No